CLINICAL TRIAL: NCT07313813
Title: A Study to Evaluate the Effect of Fasting Duration and Temporary Withholding of Dulaglutide on Retained Gastric Contents Using Gastric Ultrasound in Participants With Type 2 Diabetes Mellitus
Brief Title: A Study to Evaluate the Effect of Fasting Duration and Dulaglutide (LY2189265) Withholding on Gastric Retention in Participants With Type 2 Diabetes Mellitus
Acronym: GBGT
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 27367; H9X-MC-GBGT (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
Keywords: Point of Care Ultrasound (POCUS)
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dulaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dulaglutide (LY2189265)-Solid-Meal (Experimental): Administered subcutaneously (SC)
  Interventions: Drug: Dulaglutide
- Dulaglutide (LY2189265)-Liquid-Meal (Experimental): Administered SC
  Interventions: Drug: Dulaglutide

INTERVENTIONS:
Drug: Dulaglutide — Administered SC

SUMMARY:
The purpose of this study is to evaluate how fasting and stopping the use of Dulaglutide (LY2189265) affect the amount of food and drink that stays in your stomach after a meal.

Ultrasound devices will be used to check the stomach content after a test meal.

The study can last approximately 28 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants with Type 2 Diabetes Mellitus (T2DM) as determined by medical history and have:

  * a diagnosis of T2DM for at least 6 months
  * T2DM controlled with diet and exercise alone or are on a stable dose of metformin, with or without 1 additional oral antihyperglycemic medication, a dipeptidyl peptidase-4 (DPP-4) inhibitor or sodium glucose transporter-2 inhibitor (SGLT-2i), for at least 1 month, and
  * a hemoglobin A1c value at screening of greater than or equal to 6.5% and less than or equal to 10.0%

Exclusion Criteria:

* Have a known clinically significant gastric emptying abnormality (for example, gastroparesis or gastric outlet obstruction), have undergone weight loss surgery such as gastric bypass (bariatric) surgery or restrictive bariatric surgery (for example, Lap-Band®), or have had endoscopic and/or device-based therapy for obesity or have had device removal within the last 6 months (for example, mucosal ablation, gastric artery embolization, intragastric balloon, and duodenal-jejunal bypass sleeve)
* Have a significant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal (GI), endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs, or of constituting a risk when taking the study drug, or of interfering with the interpretation of data
* Participants who have clinical laboratory test results, blood pressure, and pulse rate that are outside the normal reference range for the population
* Have obesity induced by other endocrinologic disorders (for example, Cushing Syndrome) or diagnosed monogenetic or syndromic forms of obesity (for example, melanocortin 4 receptor deficiency or Prader-Willi Syndrome)

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-29 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of Fasting Participants with Lack of Gastric Content Retention Post-Solid Test Meal | Day 116 (at 6, 8, 12, 18 and 24 hours after baseline or Day 115 solid test meal)
  Percentage of Fasting Participants with Lack of Gastric Content Retention Post-Solid Test Meal

SECONDARY OUTCOMES:
Percentage of Fasting Participants with Lack of Gastric Content Retention After Dulaglutide (LY2189265) Post-Liquid Test Meal | Day 123 (at 6, 8, 12, 18 and 24 hours after Day 122 liquid test meal)
  Percentage of Fasting Participants with Lack of Gastric Content Retention After Dulaglutide (LY2189265) Post-Liquid Test Meal
Percentage of Fasting Participants with Lack of Gastric Content Volume Post-Liquid Test Meal After Dulaglutide (LY2189265) | Day 123 (at 6, 8, 12, 18 and 24 hours after Day 122 liquid test meal)
  Percentage of Fasting Participants with Lack of Gastric Content Volume Post-Liquid Test Meal After Dulaglutide (LY2189265)
Percentage of Fasting Participants with Lack of Gastric Content Volume Post-Solid Test Meal After Dulaglutide (LY2189265) | Day 116 (at 6, 8, 12, 18 and 24 hours after baseline or Day 115 solid test meal)
  Percentage of Fasting Participants with Lack of Gastric Content Volume Post-Solid Test Meal After Dulaglutide (LY2189265)
Percentage of Participants with Lack of Gastric Content Retention Post-Solid Test Meal After Discontinuation of Dulaglutide (LY2189265) | Baseline, through 8 days after discontinuation of dulaglutide at 6, 8, 12, 18 and 24 hours
  Percentage of Participants with Lack of Gastric Content Retention Post-Solid Test Meal After Discontinuation of Dulaglutide (LY2189265)
Percentage of Participants with Grades 0, 1, 2 from Antrum Grading Scale Post-Solid Test Meal After Dulaglutide (LY2189265) | Day 116 (at 6, 8, 12, 18 and 24 hours after baseline or Day 115 solid test meal)
  Percentage of Participants with Grades 0, 1, 2 from Antrum Grading Scale Post-Solid Test Meal After Dulaglutide (LY2189265)
Percentage of Participants with Grades 0, 1, 2 from Antrum Grading Scale Post-Liquid Test Meal After Dulaglutide (LY2189265) | Day 123 (at 6, 8, 12, 18 and 24 hours after Day 122 liquid test meal)
  Percentage of Participants with Grades 0, 1, 2 from Antrum Grading Scale Post-Liquid Test Meal After Dulaglutide (LY2189265)
Percentage of Participants with Grades 0, 1, 2 from Antrum Grading Scale Post-Solid Test Meal After Discontinuation of Dulaglutide (LY2189265) | Baseline, through 8 days after discontinuation of dulaglutide at 6, 8, 12, 18 and 24 hours
  Percentage of Participants with Grades 0, 1, 2 from Antrum Grading Scale Post-Solid Test Meal After Discontinuation of Dulaglutide (LY2189265)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Lilly Centre for Clinical Pharmacology, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Lilly Trials — https://trials.lilly.com/en-US/trial/678715